CLINICAL TRIAL: NCT05867160
Title: A 12-month, Prospective, Observational Study in Adult Patients With Focal Onset Seizures Who Are Treated With Adjunctive ASM in Real World Setting
Brief Title: Adjunctive Anti-seizure Medication (ASM) Real World Evidence (RWE) Study
Status: Active, not recruiting | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Other Study IDs: 169(A)MD21254
Record Dates: First submitted 2023-03-21; First posted 2023-05-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; Focal-onset seizure; Cenobamate; Adjunctive Therapy
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients with focal-onset seizures starting a treatment with ASM as adjunctive therapy: Adult patients having focal-onset seizures not adequately controlled despite a history of treatment with at least 2 ASM.
  The patients should be eligible to start a treatment with ASM as adjunctive therapy.The patients will be prospectively observed up to 12 months after having completed the related titration.
  Interventions: Other: ASM as adjunctive therapy

INTERVENTIONS:
Other: ASM as adjunctive therapy — ASM approved as adjunctive therapy

SUMMARY:
The purpose of this study is to describe the effectiveness of the adjunctive ASM treatment on the clinical response, safety profile and quality of life of patients affected by focal onset seizures in a real-world setting.

DETAILED DESCRIPTION:
The aim of the study is to assess the effectiveness and safety of adjunctive therapy in a real-world setting of patients affected by focal-onset seizures who are eligible to start the treatment with ASM as adjunctive therapy according to the physician's judgment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any ethnic origin ≥18 years old at baseline.
* Patients with diagnosis of focal-onset seizures with or without secondary generalization.
* Patients should have been eligible to start treatment with ASM as adjunctive therapy according to the physician's judgement prior to the inclusion.
* Patients should have clinical history of treatment failure with at least 2 ASMs.
* Patients using their seizure diary as part of their standard of care for at least 3 months prior to -the study entry (diary can be paper or electronic, filled in by patient and/or family members).
* Written informed consent (including data privacy consent) signed by the patient, legal guardian, or legally authorized representative prior to entering the study in accordance with the ICH GCP guidelines

Exclusion Criteria:

* Patients who meet any of the contraindications to the administration of adjunctive ASMs according to their approved SmPC.
* Progressive neurological disease, including degenerative CNS diseases and progressive tumors.
* Patients with unstable psychiatric diagnosis that may confound participants' ability to participate in the study or that may prevent completion of the protocol-specified assessments (e.g., in the judgement of the Investigator, pose an appreciable risk for suicide, including suicidal behavior and ideation within 6 months prior to enrollment, current psychotic disorder, acute mania).
* Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the Investigator could affect the participant's safety or interfere with study assessments.
* Patients with substance abuse or dependence (except for caffeine and nicotine).
* Patients participating in any pharmacological or nonpharmacological interventional study within 30 days prior to baseline.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with epilepsy having focal-onset seizures with or without secondary generalization not adequately controlled despite a history of treatment with at least 2 anti-seizure medications and who will meet all the inclusion and none of the exclusion study criteria.
  The patients should be eligible to start a treatment with ASM as adjunctive therapy according to the physician's judgement, that must be clearly separated from the physician's decision to include the patient in the current study. The patients will be prospectively observed up to 12 months after having completed the related titration.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in seizure frequency at 6 months of maintenance | At 6 months of maintenance compared to baseline
  The effectiveness of adjunctive ASM is measured as change in seizure frequency at 6 months of maintenance compared to baseline

SECONDARY OUTCOMES:
Change in seizure frequency at 3, 9, 12 months of maintenance | At 3, 9, 12 months of maintenance compared to baseline
  The effectiveness of adjunctive ASM is measured as change in seizure frequency at 3, 9, 12 months of maintenance compared to baseline
50, 75, 90 Percent Responder rate | At 3, 6, 9, and 12 months of maintenance phase.
  The effectiveness is measured as 50, 75, 90 Percent Responder rate
100 Percent Responder rate | At 3, 6, 9, and 12 months of maintenance phase.
  The effectiveness is measured as number/percentage of seizure free patients
Retention rate | At 3, 6, 9, and 12 months of maintenance phase.
  The effectiveness is measured as percentage of patients remaining in the study and on adjunctive therapy
Anxiety assessment | At baseline, immediately after completion of titration, at 3 months, 6 months, and 12 months of maintenance phase.
  The assessment is measured by means of the Generalized Anxiety Disorder (GAD-7) scale. Scoring GAD-7 Anxiety Severity is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety.
Depression assessment | At baseline, immediately after completion of titration, at 3 months, 6 months, and 12 months of maintenance phase.
  The assessment is measured through the Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) scale. This is a validated screening tool for depression in patients with epilepsy that consists of a 6- item questionnaire. NDDI-E scores greater than 15 were considered positive for depression, as this score was previously shown to have a specificity of 90%, sensitivity of 81%, and positive predictive value of 0.62 for a diagnosis of major depression.
Quality of life (QOL) | At baseline, immediately after completion of titration, at 3 months, 6 months, and 12 months of maintenance phase.
  The quality of life is measured by means the Quality Of Life In Epilepsy (QOLIE-31-P) questionnaire. This is a 38 questions survey of health-related quality of life for adults (18 years or older) with epilepsy. This version differs from the original QOLIE-31 (version 1) in the addition of questions about how much distress you feel about problems and worries related to epilepsy. This questionnaire should be completed only by the person who has epilepsy (not a relative or friend). Patients are asked to answer every question by circling the appropriate number (1, 2, 3...).
Cognitive assessment | At baseline, immediately after completion of titration, at 3 months, 6 months, and 12 months of maintenance phase.
  The assessment of perceived cognitive deficits is measured through the Perceived Deficits Questionnaire (PDQ-5). The PDQ-5 assesses cognitive dysfunction in people with depression. This patient-reported questionnaire includes five items measuring attention/concentration, retrospective memory, prospective memory, and planning/organization over the past four weeks. The total score ranges from 0 to 20; higher scores indicate greater perceived cognitive dysfunction.
Adverse events (AEs) | Through study completion, an average of 1 year
  Number of Adverse events (AEs) occurred (including AEs of special interest as Drug Reaction with Eosinophilia and Systemic Symptoms, rash/hypersensitivity, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico "Carlo Besta" U.O. Epilettologia Clinica e Sperimentale - Centro di Medicina del Sonno, Milan, Italy

IPD SHARING:
Plan to Share IPD: No